CLINICAL TRIAL: NCT04259034
Title: Assessment of Periodontal Status in Patients With Oral Lichen Planus
Brief Title: Periodontal Status in Oral Lichen Planus Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: RMA PGIDS/IEC/2019/32
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- systemically healthy individuals with oral lichen planus: systemically healthy individuals diagnosed with oral lichen planus on clinical and histopathological basis.
  Interventions: Other: diagnosis of periodontitis in oral lichen planus patients
- systemically healthy individuals without oral lichen planus: systemically healthy individuals without any clinical feature of oral lichen planus.
  Interventions: Other: diagnosis of periodontitis in systemically healthy individuals without oral lichen planus

INTERVENTIONS:
Other: diagnosis of periodontitis in oral lichen planus patients — diagnosis of periodontitis in oral lichen planus patients
  Groups: systemically healthy individuals with oral lichen planus
Other: diagnosis of periodontitis in systemically healthy individuals without oral lichen planus — diagnosis of periodontitis in systemically healthy individuals without oral lichen planus
  Groups: systemically healthy individuals without oral lichen planus

SUMMARY:
The aim is to investigate the influence of oral lichen planus on periodontal status of systemically healthy individuals.

DETAILED DESCRIPTION:
Lichen planus, a chronic immune-mediated inflammatory disease affects the skin and mucous membranes. Oral lichen planus is the mucosal counterpart of cutaneous lichen planus. It was reported first described in 1866 as white papular eruptions in the oral cavity. The prevalence of OLP varies from 0.1% to 4%. OLP mostly occurs in middle aged and elderly patients, with female to male ratio of 3:2. OLP is characterized by lesions consisting of radiating white, grey, velvety, thread-like papules in a linear, annular and retiform arrangement forming typical lacy, reticular patches, rings and streaks. The lesions are most common on buccal mucosa, tongue, lips, gingiva, floor of mouth, palate. Clinically OLP has six clinical presentations namely reticular, erosive, atrophic, plaque-like, papular, bullous.

Reticular form, the most common clinical form presents as fine, asymptomatic intertwined lace-like pattern called "Wickham striae" in a bilateral symmetrical form. It mainly involves the posterior mucosa of the cheek. Erosive OLP represents symptomatic lesions. Atrophic lesions may resemble the combination of two clinical forms, such as the presence of white striae characteristic of the reticular type surrounded by an erythematous area. Plaque-like form mainly found on dorsum of the tongue and the mucosa of the cheek reveals whitish homogeneous irregularities similar to leukoplakia. Papular form presents with small white papules with fine striae in its periphery. Bullous form is the most unusual clinical form, exhibiting blisters that increase in size and tend to rupture, leaving the surface ulcerated and painful.

The pathogenesis of the disease is characterized by cytotoxic CD8+ T lymphocytes migration to the epithelium inducing apoptosis of basal keratinocytes. A number of etiological factors in OLP have been proposed such as local and systemic inducers of cell-mediated hypersensitivity, drugs, dental materials, infectious agents, and stress. The existence of a local cell-mediated immune disorder has been postulated as a factor underlying development of the lesions specifically, a delayed cellular hypersensitivity response probably triggered by some exogenous agent. Periodontal diseases are the most prevalent oral microbial infections that lead to chronic inflammation of the supporting tissues of teeth. Periodontal disease has a complex pathogenesis involving host microbiome interactions. It has an impact on both local and systemic health. The pathogenesis of periodontal disease involves a local inflammatory reaction and the activation. Thus, it is possible to speculate that some interference could exist and that the potential effect arising from these shared mechanisms⁄ mediators could be localized to sites where OLP lesions are present and alteration of host immune response in OLP may have an impact on periodontal health. With this consideration, the present study is aimed to assess periodontal status in systemically healthy individuals with and without oral lichen planus.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 40-50 yrs. Clinically diagnosed and histo-pathologically confirmed cases of oral Lichen Planus

Exclusion Criteria:

History of periodontal therapy in last one year. Drug-induced lichenoid reaction or any other red or white lesions in the oral cavity.

The presence of any tooth restoration near the lesions. Smokers or patients with history of smoking. systemic diseases or conditions that are reported to be associated with periodontal diseases, including diabetes mellitus, osteoporosis, rheumatoid arthritis Pregnant and lactating women. Patients with history of systemic treatment for oral Lichen Planus Patients with cutaneous lichen planus

Ages: 40 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: systemically healthy individuals with and without oral lichen planus
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level | 6 months
  CAL will be measured from cementoenamel junction to the base of the pocket using a periodontal probe at 6 sites

SECONDARY OUTCOMES:
Bleeding on probing | 6 months
  BOP will be measured using a periodontal probe at 4 sites
PLAQUE INDEX | 6 months
  PI will be measured using a periodontal probe at 4 sites
Gingival index | 6 months
  Gingival index will be measured using a periodontal probe at 4 sites
Probing pocket depth | 6 months
  Probing pocket depth will be measured from gingival margin to the base of the pocket using a periodontal probe at 6 sites

CONTACTS AND LOCATIONS:
Overall Officials: RMA ARYA, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES, ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol